CLINICAL TRIAL: NCT05377541
Title: Comparison of PENG Block and Fascia Iliaca Compartment Block in the Postoperative Pain Control of Hip Capsular Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Carles Espinos Ramírez, Principal Investigator, Consorci Sanitari de Terrassa
Other Study IDs: 01-22-270-037
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Hip Fractures
Keywords: subcapital; hip fracture; PENG; Fascia iliaca compartment block; Postoperative pain
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PENG block: To perform the PENG block, the patient will be placed in the supine position and with the convex transducer in a transverse plane over the anteroinferior iliac spine, the probe will be aligned with the iliopectineal eminence of the pubic ramus rotating about 45º medially.
  Interventions: Procedure: Surgical treatment of femur fracture
- Fascia iliaca compartment block: To perform the iliac fascia block, the patient is placed in the supine position and with the linear transducer placed at the junction of the middle third with the lateral third of the inguinal ligament, the needle is inserted through the fascia lata and the iliac fascia.
  Interventions: Procedure: Surgical treatment of femur fracture

INTERVENTIONS:
Procedure: Surgical treatment of femur fracture — Definitive surgical treatment of femur fracture.

SUMMARY:
A prospective cohort study comparing PENG block versus iliac fascia block with the aim of evaluating its effectiveness in the peri-surgical analgesia of intracapsular femoral fracture.

DETAILED DESCRIPTION:
Hip fractures are a very common clinical situation in elderly patients and are associated with significant morbidity and mortality. In addition, they have a great social and economic impact that in most cases requires definitive surgical treatment.

Although it is a very common procedure, in proximal femur surgery there is great variability with respect to anesthetic procedures and their subsequent management. Subarachnoid anesthesia is the most commonly used for this type of surgery. During the last few years, different locoregional techniques have been described with the aim of improving perioperative analgesia in these patients. Some examples are the iliac fascia block, the 3-in-1 block or the femoral nerve block, which allow a lower consumption of opioids and reduce some adverse effects such as postoperative delirium.

The PENG (Pericapsular Nerve Group) block is a block recently described for pain management in proximal femoral surgery. It is a pure sensory block that was initially described as an analgesic technique for the treatment of acute pain after femoral fracture but has expanded its uses. Its target corresponds precisely to the described innervation of the anterior femoral capsule.

Regarding the other locoregional techniques mentioned above, these consist of non-selective blocks of the femoral, lateral femoral cutaneous and obturator nerves. Therefore, although the iliac fascia block is accepted for analgesic control of hip fracture, the PENG block is likely to be more effective because of its high selectivity.

For this reason, the investigators have decided to conduct a prospective cohort study comparing PENG block versus iliac fascia block with the aim of evaluating its effectiveness in the peri-surgical analgesia of intracapsular femoral fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subcapital, basicervical or transcervical femoral fracture in whom definitive surgical treatment is decided.
* Patients who are candidates for nerve block plus intradural anesthesia.
* Patients who agree to participate in the study

Exclusion Criteria:

* Patients with dementia or cognitive impairment (EVN not evaluable)
* Polytraumatized patient
* Patient's refusal to participate in the study
* Patient's refusal to undergo intradural anesthesia or the blockade
* Patient with sensory or motor deficits prior to surgery.
* Patient with anticoagulation or antiplatelet therapy at the time of surgery.
* Hemodynamically unstable patient or patient who becomes unstable during surgery.
* Patient allergic to the local anesthetic.
* Patient with chronic pain in treatment
* Patient with capital femur fracture

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population admitted to the hospital and scheduled for definitive surgical treatment of femur fracture.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Post-surgical pain after the disappearance of the motor block | Approximately from 1 to 2 hours after de surgery, when the effect of the spinal anesthesia disappears.
  Pain will be assessed through the Verbal Numerical Scale (VNS). The VNS is a numeric scale with a minimum value of 0 and a maximum of 10 where 0 means no pain and 10 maximum pain.
Pain 24 hours after surgery | 24 hours after surgery
  Pain will be assessed through the Verbal Numerical Scale (VNS). The VNS is a numeric scale with a minimum value of 0 and a maximum of 10 where 0 means no pain and 10 maximum pain.
Need for rescue analgesia | 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allard C, Pardo E, de la Jonquiere C, Wyniecki A, Soulier A, Faddoul A, Tsai ES, Bonnet F, Verdonk F. Comparison between femoral block and PENG block in femoral neck fractures: A cohort study. PLoS One. 2021 Jun 4;16(6):e0252716. doi: 10.1371/journal.pone.0252716. eCollection 2021. PMID 34086782
- [Background] Jadon A, Mohsin K, Sahoo RK, Chakraborty S, Sinha N, Bakshi A. Comparison of supra-inguinal fascia iliaca versus pericapsular nerve block for ease of positioning during spinal anaesthesia: A randomised double-blinded trial. Indian J Anaesth. 2021 Aug;65(8):572-578. doi: 10.4103/ija.ija_417_21. Epub 2021 Aug 25. PMID 34584279
- [Background] Acharya U, Lamsal R. Pericapsular Nerve Group Block: An Excellent Option for Analgesia for Positional Pain in Hip Fractures. Case Rep Anesthesiol. 2020 Mar 12;2020:1830136. doi: 10.1155/2020/1830136. eCollection 2020. PMID 32231802
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experiences of pericapsular nerve group (PENG) block for hip surgery. J Clin Anesth. 2018 Dec;51:60-61. doi: 10.1016/j.jclinane.2018.08.003. Epub 2018 Aug 8. No abstract available. PMID 30096522 (Retraction: PMID 35393178 J Clin Anesth. 2022 Aug;79:110722)
- [Background] Sahoo RK, Jadon A, Sharma SK, Peng PW. Peri-capsular nerve group block provides excellent analgesia in hip fractures and positioning for spinal anaesthesia: A prospective cohort study. Indian J Anaesth. 2020 Oct;64(10):898-900. doi: 10.4103/ija.IJA_450_20. Epub 2020 Oct 1. No abstract available. PMID 33437080
- [Derived] Esteller PG, Ramirez CE, Juarez-Pomes M, Martin Sanchez JC, Martinez Garcia M. PENG Block: A superior alternative for pain management in intracapsular hip fractures. Saudi J Anaesth. 2025 Apr-Jun;19(2):251-256. doi: 10.4103/sja.sja_96_25. Epub 2025 Mar 25. PMID 40255360